CLINICAL TRIAL: NCT04143503
Title: Observational Cohort Study to Characterise the Current Use of Parenteral Nutrition and Clinical Outcomes in Adult Critically Ill Patients Hospitalised in Intensive Care Units in Europe
Brief Title: Observational Cohort Study on the Use of Parenteral Nutrition and Clinical Outcomes in Adult Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Collaborators: IQVIA Commercial GmbH & Co. OHG (Industry)
Responsible Party: Sponsor
Other Study IDs: NScr-003-CNI
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Critical Illness
Keywords: ICU; parenteral nutrition; enteral nutrition; energy intake; protein intake
MeSH Terms: conditions — Critical Illness; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult critically ill patients

SUMMARY:
The aim of this study is to characterise the use of clinical nutrition support, especially of parenteral nutrition that is administered directly into a vein, in adult patients with critical illness. The study wants to assess nutritional balance (that means the ratio of calories and protein prescribed to calories and protein actually received). Furthermore, it wants to evaluate whether the nutrition received has influence on the patients' clinical outcome, with focus on measures of physical function, such as capability of conducting daily living activities. As the study is "observational", no specific medications or treatments will be provided as part of the study to the patients.

Study patients will be observed during their stay on an intensive care unit, for a maximum duration of 15 days. Furthermore, questions on the well-being of the patients will be asked via telephone interviews 30 and 90 days after their admission to the intensive care unit.

Data of approximately 1250 patients will be collected and evaluated in this study, from approximately 100 hospitals in 11 European countries (Austria, Belgium, Czech Republic, France, Germany, Hungary, Italy, Poland, Spain, Sweden and United Kingdom).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤95 years, male or female
2. Hospitalised in a medical, surgical, or trauma ICU for at least five consecutive calendar days and either admitted to the ICU during the predefined screening month or admitted to the ICU maximally 4 days before start of the screening month
3. BMI ≥18.5 kg/m2 and ≤45 kg/m2
4. Written informed consent or requirements of local/national ethical committee

Exclusion Criteria:

1. Burn injury
2. Pre-existing neuromuscular or psychiatric disorders that preclude proper assessment of functional status
3. Severe hypoxic brain injury or severe neurological diagnosis (e.g. meningitis, encephalitis, brain trauma, spinal cord injury) at the time of ICU admission that precludes proper assessment of functional status
4. Receiving home parenteral nutrition at the time of ICU admission (e.g. due to short bowel syndrome)
5. Receiving home enteral nutrition (tube feeding) at the time of ICU admission
6. Chronic invasive or chronic non-invasive ventilatory support before ICU admission
7. Patients with a legal representative in place before ICU admission
8. Admission to the ICU for palliative care
9. Previous participation in this study (if the screening month is repeated and a patient is re-admitted to the ICU during the repeated screening month, only ICU data collected for that patient during the original screening month will be included)
10. Concurrent enrolment in a nutrition-related interventional study at the time of screening

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult male and female patients with critical illness (i.e. patients requiring pharmacological and/or technical support to treat a vital threat) who are hospitalised in a medical, surgical, or trauma ICU for at least 5 consecutive calendar days.
Sampling Method: Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving enteral nutrition (EN), parenteral nutrition (PN), and oral nutrition (ON)/oral nutrition supplements (ONS) | from admission to ICU until discharge from ICU or death (maximum of 15 days)
Cumulative caloric balance | from admission to ICU until discharge from ICU or death (maximum of 15 days)
Cumulative protein balance | from admission to ICU until discharge from ICU or death (maximum of 15 days)
Cumulative calories (kcal/kg and total kcal) administered via EN, PN, ON/ONS, and concomitant medications (e.g. propofol, glucose, citrate, clevidipine), and via all sources combined | from admission to ICU until discharge from ICU or death (maximum of 15 days)
Cumulative protein (g/kg and total g) administered via EN, PN, ON/ONS, and via all sources combined | from admission to ICU until discharge from ICU or death (maximum of 15 days)
Proportion of patients with interrupted/stopped or not started clinical nutrition | from admission to ICU until discharge from ICU or death (maximum of 15 days)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hiesmayr, Prof. MD, Principal Investigator — Medical University of Vienna
Locations (76):
- Medical University of Vienna, Vienna, Austria
- Belgium (9):
  - Vivalia - Clinique Saint Joseph, Arlon
  - Hospital Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Clinique Universitaire Saint-Luc - Université Catholique de Louvain (UCL), Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - University Hospital Antwerp, Edegem
  - Ghent University Hospital, Ghent
  - Saint-Pierre Clinic, Ottignies
  - Hospital Center of Wallonie Picarde, Tournai
- Czechia (13):
  - Clinic of Anesthesiology, Resuscitation and Intensive Care, University Hospital Brno, Brno
  - Clinic of Internal Medicine and Gastroenterology, University Hospital Brno, Brno
  - St Anne's University Hospital Brno, Brno
  - 3rd Department of Internal Medicine - Metabolic Care and Gerontology, University Hospital Hradec Králové, Hradec Králové
  - Clinic of Anesthesiology, Resuscitation and Intensive Care, University Hospital Hradec Králové, Hradec Králové
  - III Internal Gerontometabolic Clinic, University Hospital Hradec Králové, Hradec Králové
  - University Hospital Olomouc Palacky University in Olomouc Faculty of Medicine and Dentistry, Olomouc
  - Hospital Pardubice Region, Inc., Pardubice
  - Charles University Hospital Plzen, Pilsen
  - University Hospital Pilsen University Hospital in Pilsen (Fakultní nemocnice Plzeň: Úvodní strana), Pilsen
  - General University Hospital Prague, Prague
  - Motol University Hospital, Prague
  - Masaryk Hospital, Ústí nad Labem
- France (13):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Hôpital de la Cavale Blanche à Brest, Brest
  - Hospital Center University of Caen Normandie, Caen
  - Hôpital Trousseau - Surgical Intensive Care Unit, Chambray-lès-Tours
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Grenoble - Hôpital Michallon, La Tronche
  - Hospices Civils de Lyon - Hópital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire de Saint-Étienne - Hopital Nord, Saint-Etienne
  - Hôpital Foch, Suresnes
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Charité Universitätsmedizin - Campus Benjamin Franklin, Berlin
  - Charité Universitatsmedizin - Medizinische Klinik mit Schwerpunkt Nephrologie und Internistische Intensivmedizin, Berlin
  - Augusta Kliniken Bochum Hattingen, Bochum
  - KRH Klinikum Siloah - Klinik für Gastroenterologie, Interventionelle Endoskopie und Diabetologie, Hanover
  - UKSH Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Klinikum St. Georg, Leipzig
  - Klinikum der Universität München, Munich
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Klinikum Wetzlar-Braunfels - Klinik für Geriatrie, Wetzlar
- Hungary (6):
  - Dél-Pesti Centrumkórház - National Institute of Hematology and Infectiology, Budapest
  - MH EK Honvédkorház, Budapest
  - University of Debrecen - Department of Anaesthesiology and Intensive Therapy, Debrecen
  - Jósa András Oktatókórház, Nyíregyháza
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár
  - Csolnoky Ferenc Kórház, Veszprém
- Italy (5):
  - Ospedali Riuniti di Foggia, Foggia
  - Ospedale San Paolo, Milan
  - Ospedale Umberto I, Nocera Inferiore
  - Hospital Santa Maria delle Croci, Ravenna
  - Ospedale Infermi Rimini, Rimini
- Poland (6):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - 10 Wojskowy Szpital Kliniczny z Polikliniką w Bydgoszczy, Bydgoszcz
  - Medical University of Silesia, Katowice
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie sp. Z o.o., Krakow
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Szpital Wojewódzki w Poznaniu, Poznan
- Spain (10):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Dr Josep Trueta de Girona - Intensive Care Unit, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario de Fuenlabrada - Intensive Care Unit, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Clinic de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Alvaro Cunqueiro, Vigo
- Karolinska University Hospital, PMI Huddinge, B31, Stockholm, Sweden
- United Kingdom (3):
  - Liverpool Heart and Chest Hospital, Liverpool
  - The Royal Liverpool University Hospital, Liverpool
  - The Royal London Hospital, Barts Health NHS Trust & Queen Mary University of London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matejovic M, Huet O, Dams K, Elke G, Vaquerizo Alonso C, Csomos A, Krzych LJ, Tetamo R, Puthucheary Z, Rooyackers O, Tjader I, Kuechenhoff H, Hartl WH, Hiesmayr M. Medical nutrition therapy and clinical outcomes in critically ill adults: a European multinational, prospective observational cohort study (EuroPN). Crit Care. 2022 May 18;26(1):143. doi: 10.1186/s13054-022-03997-z. PMID 35585554
- [Derived] Hiesmayr M, Csomos A, Dams K, Elke G, Hartl W, Huet O, Krzych LJ, Kuechenhoff H, Matejovic M, Puthucheary ZA, Rooyackers O, Tetamo R, Tjader I, Vaquerizo C. Protocol for a prospective cohort study on the use of clinical nutrition and assessment of long-term clinical and functional outcomes in critically ill adult patients. Clin Nutr ESPEN. 2021 Jun;43:104-110. doi: 10.1016/j.clnesp.2021.01.048. Epub 2021 Feb 12. PMID 34024501